CLINICAL TRIAL: NCT07386886
Title: A Multicenter Cohort Study of Leptomeningeal Metastasis in Breast Cancer: Clinical Characterization and Development of a Novel Graded Prognostic Assessment (BC-LGPA) Model
Brief Title: Development of a Novel Graded Prognostic Assessment (BC-LGPA) Model for Breast Cancer Leptomeningeal Metastasis
Status: Completed | Type: Observational
Sponsor: Jian Zhang,MD (Other)
Responsible Party: Sponsor-Investigator, Jian Zhang,MD, Director of Phase I clinical Research ward, Fudan University
Organization: Fudan University (Other)
Other Study IDs: 260126
Record Dates: First submitted 2026-01-26; First posted 2026-02-04 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Leptomeningeal Metastasis in Breast Cancer

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: systematic therapy — Patients with BCLM receive systematic therapy，IT and radiation.

SUMMARY:
The investigators conducted a large, multicenter retrospective study of patients with breast cancer leptomeningeal metastasis (BCLM), constituting one of the largest and most comprehensively curated cohorts to date. Data from 403 patients diagnosed between November 2013 and November 2025 were collected from three major academic centers. Detailed clinical, pathological, diagnostic, and treatment data were analyzed. Overall survival (OS) was evaluated, and independent prognostic factors were identified via Cox regression. A novel Breast Cancer Leptomeningeal Graded Prognostic Assessment (BC-LGPA) model was developed and validated for risk stratification.

ELIGIBILITY:
Inclusion Criteria:

* patients with BCLM

Exclusion Criteria:

* patients with other BC CNS metastasis

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: The investigators conducted a large, multicenter retrospective study of patients with breast cancer leptomeningeal metastasis (BCLM), constituting one of the largest and most comprehensively curated cohorts to date. Data from 403 patients diagnosed between November 2013 and November 2025 were collected from three major academic centers.
Sampling Method: Non-Probability Sample
Enrollment: 403 (Actual)
Dates: Start 2013-11-30 (Actual); Primary Completion 2025-11-30 (Actual); Study Completion 2026-01-26 (Actual)

PRIMARY OUTCOMES:
Overall survival | Up to approximately 30 months
  Time from date of randomization to the date of death from any cause